CLINICAL TRIAL: NCT05476289
Title: Effect of a Partially Hydrolyzed Formula with Added Synbiotics on Growth and Immune-related Outcomes in Chinese Children Up to Four Years of Age: a Follow-up Study of a Clinical Trial in the First Year of Life
Brief Title: A Follow-up Study of Dragon Study (NCT03520764): to Assess the Growth and Immune-related Outcomes
Status: Completed | Type: Observational
Sponsor: Danone Nutricia (Industry)
Collaborators: Nutricia Early Life Nutrition (Shanghai) Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: ELNCN2204
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool Sample will be retained on Baseline visit and Visit 4 (48months)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- A: children who received partially hydrolyzed formula containing synbiotics in the first 17 weeks of life in the Dragon study.
  Interventions: Other: No intervention
- B: children who received standard infant formula containing prebiotics in the first 17 weeks of life in the Dragon study.
  Interventions: Other: No intervention
- C: children who received full breastfeeding in the first 17 weeks of life in the Dragon study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Dragon follow-up aims to evaluate the growth, allergies, and infections of Chinese subjects up to four years of age who completed the intervention period visit (from Day 0-44 to Week 17) of the Dragon study [EBB16SI08406]. This study aims to provide insights into the role of usage of a partially hydrolyzed formula with added synbiotics in early life children's growth and immune-related outcome up to 4 years of age.

DETAILED DESCRIPTION:
After providing informed consent, subjects from the prior randomized controlled trial (Dragon study) will be enrolled in the follow-up study. The observation period is from the end of the Dragon study (12 months) to 4 years of age. Data from the end of the Dragon study to the actual age at the enrolment (with 4 years of age as the upper limit) will be collected retrospectively, and data from the actual age at the enrolment (if younger than 4 years of age) to 4 years of age will be collected prospectively. Data will be collected retrospectively or prospectively at four scheduled visit timepoints: 24 months, 30 months, 3 years and 4 years of age. The visit points are in accordance with the health assessment schedule of the Maternal and Children Health Network in China to ensure the data on growth before the start of this follow-up study is available.

As required by relevant law issued by the National Health and Family Planning Commission in China, the maternal and children health network institutions in all provinces should carry out regular health assessments for children aged 0-6 years, in which the growth evaluations should be conducted for children aged 24 months, 30 months, 3 years and 4 years. In this follow-up study, the weight and height parameters will be obtained from the Children's Health Manual, and skinfolds thickness at 4 years of age will be measured on-site by trained personnel.

Except for stool microbiota collection and skinfold thickness measurement, all variables will be collected via our online tools. Data on growth parameters, allergy, infection, medications, and hospitalization will be collected using an electronic data capture system (EDC). Parents are expected to login to an electronic platform at a scheduled time from an Internet-accessible smartphone or tablet to fill the online questionnaire and send photocopies of examination results as required (any information related to personal privacy such as name, address and hospitalization ID should be covered before being taken a photocopy, see section 11.5). Parents will receive reminder short messages on the first day of the scheduled visit window. Those who fail to respond to the follow-up message in two weeks will receive a backup telephone call to complete the filling.

The gastrointestinal symptoms, stool assessment, skinfold thickness and dietary pattern and behaviour will only be collected prospectively. If the subjects' actual age at the enrolment is older than 4 year old, skinfolds thickness, gastrointestinal symptoms, stool assessment and dietary pattern and behaviour at 4 years of age will not be collected.

ELIGIBILITY:
Inclusion Criteria:

* Children completed the intervention period visits (from Day 0-44 to Week 17) of the Dragon study in one of the randomized groups or in the breastfeeding reference group.
* Children whose parents provide informed consent for participation in the Dragon Follow Up study.

Exclusion Criteria:

* Participated or currently in another interventional clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of healthy term-born children who completed the intervention period visit (from Day 0-44 to Week 17) of the preceding Dragon study, irrespective of whether they participated in one of the randomised groups or in the breastfeeding reference group. In total, 226 subjects had completed the Week 17 visit in the Dragon study. The subjects will be enrolled in the Dragon follow up after obtaining informed consent from their parents for the follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Growth | 12-month to 4-year age
  * Weight, weight gain, height, Body Mass Index (BMI) at 24 months, 30 months, 3 years and 4 years of age
  * Skin folds thickness at 4 years of age
    * Individual skin folds thickness (triceps, biceps, subscapular, suprailiac)
    * Sum of all 4 skin folds thickness
    * Subcutaneous trunk fat (sum of subscapular and suprailiac skinfolds)
    * Subcutaneous peripheral fat (sum of triceps and biceps)
  * Z-score of the following anthropometric parameters up to 4 years of age according to World Health Organization (WHO) growth chart:
    * Height-for-age
    * Weight-for-age
    * BMI-for-age
    * Weight-for-height
    * Subscapular skinfold-for-age
    * Triceps skinfold-for-age
Allergy | 12-month to 4-year age
  • The occurrence of parent reported allergic manifestations and doctor diagnosed allergies (as reported by parents and noted in the subject's medical dossier) at 24 months, 30 months, 3 years and 4 years of age.
  * Respiratory: Wheeze and asthma
  * Skin: Eczema, atopic dermatitis, urticaria
  * Food: Adverse reactions to foods and food allergy (the types of foods that result in allergy should be recorded)
  * Other: Rhinitis (allergic responses to pollen, house dust mite)
Infections | 12-month to 4-year age
  • The occurrence of parent-reported infections symptoms and doctor diagnosed infections (as reported by parents and noted in the subject's medical dossier) at 24 months, 30 months, 3 years and 4 years of age. In particular,
  * Fever
  * Respiratory infections; upper respiratory tract infections, nasopharyngitis, bronchitis/bronchiolitis, pneumonia)
  * Ear infections
  * Skin infections; dermatitis
  * GI infections
Stool microbiota | 3-year age to 4-year age
  Stool microbiota at the enrolment and 4 years of age
Gastrointestinal symptoms | 12-month to 4-year age
  • The occurrence of any gastrointestinal discomfort symptoms in the past 4 weeks, including vomiting, abdominal pain, constipation, diarrhea at the enrolment and 4 years of age.
Medications | 12-month to 4-year age
  * The use of medications and/or a medical device (inhaler) to prevent or relieve allergic manifestations and allergies or infections (as reported by parents and/or noted in the subject's medical dossier).
  * Probiotics and other nutritional supplements
Hospitalisation | 12-month to 4-year age
  * Number of days hospitalised for allergic manifestations, allergies or infections (reported by parents and/or noted in the subject's medical dossier).
  * Number of visits to the emergency room, outpatient departments or clinics for allergic manifestations, allergies and infections.
Parental outcomes | 12-month to 4-year age
  • Parental loss of productive working days due to the child's allergic manifestations, allergies or infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No